CLINICAL TRIAL: NCT04088214
Title: Case Series Regarding the Efficacy of the Arthroscopic Assisted Lateral Soft Tissue Release for Hallux Valgus
Brief Title: Arthroscopic Assisted Lateral Soft Tissue Release for Hallux Valgus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTEC-2019-0340
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Hallux Valgus; Hallux Valgus and Bunion
Keywords: Arthroscopy
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Intervention Model Description: case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ArtDSTP (Experimental): Arthroscopic lateral soft tissue release
  Interventions: Procedure: Arthroscopic lateral soft tissue release

INTERVENTIONS:
Procedure: Arthroscopic lateral soft tissue release — The arthroscopic lateral soft tissue release is performed using an inside-out approach via the 1MTPJ arthroscopy.

SUMMARY:
Lateral soft tissue release is commonly performed as part of the surgical correction of hallux valgus. This study will look at the results form a series of patients whom have underwent the arthroscopic lateral soft tissue release.

ELIGIBILITY:
Inclusion:

* >18 and legally fit for consent
* Symptomatic hallux valgus with HVA >15 degrees

Exclusion:

* Active physical or mental disorders that could affect rehabilitation including

  * Other conditions affecting ambulation: lower limb injury, neuromuscular problems etc.
  * Mental incapacitation
* Previous hallux valgus surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
HVA | 12 weeks post-surgery
  • Hallux valgus angle (HVA) measured on a weight-bearing DP radiograph
HVA | 52 weeks post-surgery
  • Hallux valgus angle (HVA) measured on a weight-bearing DP radiograph

CONTACTS AND LOCATIONS:
Overall Officials: Samuel KK Ling, MBChB, Principal Investigator — Assistant Professor
Locations (1):
- CUHK, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No